CLINICAL TRIAL: NCT01598649
Title: Influence of Intervention With Lupin Protein-enriched Foods on Cardiovascular Risk Factors in Hypercholesterolemic Subjects
Brief Title: Intervention With Lupin Protein-enriched Foods in Hypercholesterolemic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil., University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H52-12
Record Dates: First submitted 2012-05-09; First posted 2012-05-15 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Hypercholesterolemia
Keywords: Dietary protein; Lupin protein; Cholesterol metabolism; Protein metabolism; Hypercholesterolemia; Protein-enriched foods
MeSH Terms: conditions — Hypercholesterolemia | interventions — Mannitol; Arginine; Milk Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lupin protein (Experimental): Lupin protein isolate (cultivar: Lupinus angustifolius Boregine; incorporated in study products) and placebo capsules with mannitol
  Interventions: Dietary Supplement: Fabricated foods with lupin protein; Dietary Supplement: Mannitol
- Milk protein (Active Comparator): Milk Protein Isolate (75% sodium caseinate (EM7; DMV international) and 25% whey protein (Megglosat HP; Meggle), incorporated in study products) and Placebo capsules
  Interventions: Dietary Supplement: Mannitol; Dietary Supplement: Fabricated foods with milk protein
- Milk protein and arginine (Active Comparator): Milk Protein Isoalte (75% sodium caseinate (EM7; DMV international) and 25% whey protein (Megglosat HP; Meggle), incorporated in study products) and 1,6 g Arginin in four caspules per day
  Interventions: Dietary Supplement: Arginine; Dietary Supplement: Fabricated foods with milk protein

INTERVENTIONS:
Dietary Supplement: Fabricated foods with lupin protein — - Foods containing altogether 25 g lupin protein isolate (bread, roll, sausage, spread)
  Arms: Lupin protein
Dietary Supplement: Mannitol — - Placebo capsules containing mannitol (four capsules per day)
  Arms: Lupin protein; Milk protein
Dietary Supplement: Arginine — - Capsules containing arginine (four capsules per day with a total daily dosage of 1,6 g)
  Arms: Milk protein and arginine
Dietary Supplement: Fabricated foods with milk protein — Foods containing altogether 25 g milk protein isolate (bread, roll, sausage, spread)
  Arms: Milk protein; Milk protein and arginine

SUMMARY:
The objective of the study is to elucidate the effects of lupin protein (Lupinus angustifolius Boregine) as part of a mixed diet on cardiovascular risk factors and to clarify the role of arginine, one of the most abundant amino acids in lupin protein.

DETAILED DESCRIPTION:
The study is based on a previous finding that a daily dosage of 25 g lupin protein isolate, administered as protein drinks, is capable to influence the plasma lipids positively.

Consequently, the physiological effects of a mixed diet containing 25 g lupin protein isolate per day will be investigated compared to 1) a diet containing 25 g of milk protein as well as to 2) a diet with 25 g milk protein and additionally the amino acid arginine supplemented daily.

A double-blinded, controlled, randomized cross-over trial will be performed. Altogether 75 volunteers with hypercholesterolemia will be divided into three groups of 25 subjects each. After a run-in period (baseline), the first group will consume foods with lupin protein isolate (group A), the second group will receive the same foods with milk protein isolate (group B) and the third group will consume the foods with milk protein and 1,6 g arginine per day over a period of four weeks. After a wash-out period of six weeks, the diet will be crossed within the three groups for a second intervention period of four weeks. After another wash-out period, diet will be crossed within the three groups once again.

Arginine will be provided as capsule (1,6 g per day = four capsules per day) in one of the two groups receiving foods with milk protein. In the other groups (receiving foods with lupin protein or milk protein only) four placebo capsules will be served, containing mannitol.

ELIGIBILITY:
Inclusion Criteria:

* Moderate Hypercholesterolemia (total cholesterol >= 5.2 mmol/L)
* Age: 20-80 years

Exclusion Criteria:

* Intake of lipid-lowering pharmaceuticals
* Allergy against legumes
* Intolerance or allergy against milk
* Pregnancy, lactation
* Chronic bowel diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in cholesterol metabolism | After 0, 4, 10, 14, 20, and 24 weeks
  Blood lipids (total cholesterol, LDL cholesterol, HDL cholesterol, cholesterol, triacylglyceroles)

SECONDARY OUTCOMES:
Changes in protein metabolism | After 0,4, 10, 14, 20, and 24 weeks
  Plasma: amino acids, total protein, albumin, urea
Changes in body composition (body status) | After 0, 4, 10, 14, 20, and 24 weeks
  Bioelectrical impedance analysis, body weight, blood pressure
Changes in high-sensitive CRP | After 0, 4, 10, 14, 20, and 24 weeks
  Inflammation marker
Changes in parameter of diabetes mellitus | After 0, 4, 10, 14, 20, and 24 weeks
  Fasting glucose

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutritional Physiology
Locations (1):
- Friedrich Schiller University Jena, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Bahr M, Fechner A, Kiehntopf M, Jahreis G. Consuming a mixed diet enriched with lupin protein beneficially affects plasma lipids in hypercholesterolemic subjects: a randomized controlled trial. Clin Nutr. 2015 Feb;34(1):7-14. doi: 10.1016/j.clnu.2014.03.008. Epub 2014 Apr 1. PMID 24746974